CLINICAL TRIAL: NCT04189107
Title: An Investigation of Postoperative Pain, Why Still in Hospital and Days Alive and Out of Hospital Following Transoral Robotic Surgery for Squamous Cell Carcinoma of Unknown Primary and Obstructive Sleep Apnea
Brief Title: Postoperative Pain, Why Still in Hospital and DAOH Following TORS for SCCUP & OSAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Candys Foundation (Unknown); Region Capital Denmark (Other); Odense University Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Mikkel Hjordt Holm Larsen, Coordinating investigator, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DexaCup
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Analgesia; Surgery; Cancer of Head and Neck; Oropharyngeal Cancer; Carcinoma of Unknown Primary; Pain, Postoperative; Postoperative Pain
MeSH Terms: conditions — Agnosia; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Neoplasms, Unknown Primary; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization to either experimental or control treatment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): High dose Dexamethasone
  Interventions: Drug: Dexamethasone
- Control (Placebo Comparator): Standard dexamethasone dosage and placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — High-dose dexamethasone peroperative and postoperative on day 2 and 4
  Other Names: High-dose
  Arms: Experimental
Drug: Placebo — low dose dexamethasone peroperative and placebo postoperatively on day 2 and 4
  Other Names: Low-dose dexamethasone
  Arms: Control

SUMMARY:
This protocol investigates the effect of a high dose dexamethasone regimen in the treatment of postoperative pain following Transoral Robotic Surgery (TORS). The protocol consists of three substudies.

1. Randomized double-blinded clinical trial assigning half of the participants to a high-dose dexamethasone regimen while the other half will receive a low-dose dexamethasone dosage and placebo in the first postoperative period.
2. A investigation of "Why in hospital?" following TORS. From the first postoperative day until discharge reasons for continued hospitalization will be registered in order to identify clinical and organizational factors contributing to hospitalization
3. An assessment of "Days Alive and Out of Hospital" following TORS. From the day of surgery and the first 12 postoperative months all admissions to a hospital ward will be registered along with admission reasons. Any death during the first 12 months will be noted with a cause of death.

DETAILED DESCRIPTION:
The morbidity after TORS has not yet been fully investigated, but a recent studies suggest that pain is one of the primary causes for unplanned readmission This issue has been investigated by Clayburgh D et al who found that a prolonged dexamethasone regime lowered the pain scores on day three after surgery. The patients treated with the prolonged dexamethasone regime also showed a significant improvement in the food consistency they were capable to swallow and had a shortened length of stay (LOS). Recently, a pilot-study showed, that an intensified dexamethasone regime among TORS patients reduced the pain level to that of a standard tonsillectomy. Besides an analgesic effect glucocorticoids furthermore poses an anti-inflammatory quality which can be used to lower the physiological stress and inflammatory response following surgery and may prevent organ dysfunctions and complications The analgesic effect of dexamethasone has been the topic of many clinical studies, and are well described in various surgical fields. However, the optimal dose and regime for glucocorticoids prescription has so far not been established. The evidence favoring one dosage regime and an optimal prescribed dose is restricted by the variance in the regimes used in various clinical trials and the fact that there is a need for clinical trial investigating steroids with pain as the primary endpoint Consequently, it is important to thoroughly investigate and optimize the analgesic regime after TORS.

Hospitalization So far when evaluating the long-term consequences of TORS, the main focus has been on oncological outcomes and quality of life with attention to functional outcomes, i.e. feeding tube dependency and dysphagia while the LOS following TORS and why the patient is hospitalized after the procedure have been sparsely studied.

The reason why TORS patients are still hospitalized after the procedure and which clinical and organizational factors contribute to the hospitalization have not yet been examined and understood but is highly relevant in order to understand and improve the postoperative care.

A method to assess the efficiency of a therapy have emerged from the cardiology field and is called Days Alive and Out of Hospital (DAOH). This has been used in investigations of heart failure patients and myocardial infarction patients. This outcome combines mortality and morbidity, and accounts for the number but also duration of several hospitalizations after the primary discharge.

DAOH has only sparse been used in the surgical field, and only in few studies in the cardiac surgery area. The measurement is a patient-centered outcome that provide better information to the patient and surgeon when planning surgery, and can be used for quality improvement studies since it accounts for effective and efficient care.

Therefore, the DAOH measurement applied to the evaluation of TORS treatment for SCCUP will benefit the insight in how the patient's life after treatment is affected.

The aims of this study comprising patients treated with TORS for SCCUP:

1. To lower the patients pain intensity after the TORS procedure with an intensified dexamethasone regimen.
2. To investigate the clinical and organizational factors contributing to hospitalization after TORS, and with this knowledge to establish an optimized postoperative care program.
3. To measure the efficiency and morbidity after TORS using DAOH as a descriptive assessment 12 months postoperatively.

This project consists of four studies:

Study 1 - Corresponding to aim A. The investigators hypothesize that an intensified dexamethasone regime will lower patients' reported pain intensity following TORS. This will be investigated in a randomized (1:1) double-blinded clinical trial among SCCUP patients undergoing TORS and extrapolated to the entire TORS population.

* A routine surgical complications study will be performed and examine surgical complications within the first 30 postoperative days.

Study 2 - Corresponding to aim B The investigators hypothesize that not much is known about the precise reasons for why patients are hospitalized following TORS. Hence, a prospective observational study regarding "why still in hospital after TORS?" will be conducted among all patients with SCCUP scheduled for TORS.

Study 3 - Corresponding to aim C The investigators hypothesize that TORS is an efficient procedure with a low morbidity. Hence, a prospective observational study regarding DAOH will be conducted among all SCCUP patients scheduled for TORS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Ability to provide a written informed consent
* ECOG/WHO performance status 0-2
* Squamous cell carcinoma of unknown primary or obstructive sleep apnea
* Booked for TORS based on radiologic and clinical assessment by an ENT surgeon oTORS for obstructive sleep apnea must be preceded by a Drug-induced sleep endoscopy (DISE) examination
* Negative Urine HCG pregnancy test for women in the fertile age.

Exclusion Criteria:

* Serious medical comorbidities (ECOG/WHO performance status >2). Other contraindications to surgery
* Distant metastasis
* Active Herpes zoster
* Previous head and neck cancer
* Significant trismus, maximum inter-incisal opening 35mm
* Insulin dependent diabetes
* Allergy to glucocorticoids
* Preoperative daily use of systemic glucocorticoids <90 days before the surgery Glucocorticoids administered to the patient's routine examination under general anesthesia with bilateral biopsies from base of the tongue, adenoidectomy and concurrent tonsillectomy are not a part of this exclusion criteria. Only systemic daily use <90 prior TORS is an exclusion criterion.
* Preoperative use of biological anti-inflammatory medication <90 days before the surgery
* Active gastric ulcer in the opinion of the investigator
* Pregnancy/Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
Patient-reported Pain intensity | Postoperative day 1 until day 14 postoperatively
  Visual analog scale (VAS) ranging from 0-10. 0 being no pain and 10 being maximum pain. The patient will twice daily self-assess pain-intensity during both rest and activity (swallowing). The pain-intensity will be noted in a pain-diary

OTHER OUTCOMES:
Why in hospital | Postoperative day 1 until discharge
  A functional discharge criteria scheme will be used twice daily at 9 a.m. and 2 p.m. (± 2 hours) to decide whether the patient can be discharged. The scheme will be filled out by a doctor and/or nurse and used until discharge from the ward. This is an assessment of organizational and clinical factors contributing to hospitalization
Days Alive and Out of Hospital | From the day of surgery and the first 12 postoperative months
  Days alive and out of hospital is a composite patient-centered endpoint. It is calculated by deducting the length of stay of the initial admission as well as any subsequently admissions and days after potential death from the total follow-up period. Days Alive and Out of Hospital will be investigated from the day of surgery with a 12 months follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology, Head and Neck Surgery & Audiology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No